CLINICAL TRIAL: NCT05411692
Title: Effects of Functional Electrical Stimulations With and Without Motor Priming Exercises on Tenodesis Grip in Patients With Spinal Cord Injury
Brief Title: Functional Electrical Stimulations With and Without Motor Priming Exercises in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0214
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Functional electrical stimulations and motor priming exercise (Experimental): Functional electrical stimulations and motor priming exercise • Palmar Grasp (holding a ball) of Lateral Grasp (holding a tray),Tripod grip (thumb, index, and middle finger: holding a pen), Two finger opposition (thumb and index finger: holding a peg, Lateral Pinch (thumb and index finger: holding a credit card), lateral pinch, two fingers (index and middle finger: smoker's grip
  Interventions: Other: Functional electrical stimulations and motor priming exercise
- Functional electrical stimulations (Active Comparator): Stimulation parameters are (1) balanced, biphasic, current-regulated electrical pulses; (2) pulse amplitude from 8 to 50 mA (typical values 17- 26 mA); (3) pulse width 250 ms; and (4) pulse frequency from 20 to 70 Hz (18). Trancutaneous stimulation will be delivered bilaterally with surface electrodes placed on the volar aspect of each wrist targeting the distribution of the median nerve
  Interventions: Other: Functional electrical stimulations
- Convetional phyusical therapy (Placebo Comparator): The prescription of resistance load for strength training will be performed with fine motor exercise , based on sub maximal repetitions
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Functional electrical stimulations and motor priming exercise — One pair of surface stimulation electrodes is placed on the subject's skin above the flexor digitorum superficialis and the flexor digitorum profundus muscles to generate finger flexion. The Second pair of electrodes is placed on the subject's skin, above the median
  nerve, to generate thumb flexion. The third pair of electrodes is placed on the subject's skin, above the extensor digitorum muscle, to generate finger extension. Motor priming exercises will be done (functional task practice, FTP) for 20 minutes. Participants will be asked to spend at least 20 minutesDuration of training will be 4 weeks, 5 days per week, one session per day, and one hour per session.
  Arms: Functional electrical stimulations and motor priming exercise
Other: Functional electrical stimulations — Stimulation parameters are (1) balanced, biphasic, current-regulated electrical pulses; (2) pulse amplitude from 8 to 50 mA (typical values 17- 26 mA); (3) pulse width 250 ms; and (4) pulse frequency from 20 to 70 Hz (18). Trancutaneous stimulation will be delivered bilaterally with surface electrodes placed on the volar aspect of each wrist targeting the distribution of the median nerve. One pair of surface stimulation electrodes is placed on the subject's skin above the flexor digitorum superficialis and the flexor digitorum profundus muscles to generate finger flexion. The Second pair of electrodes is placed on the subject's skin, above the median
  nerve, to generate thumb flexion for 20 minutes
  Arms: Functional electrical stimulations
Other: Conventional physical therapy — a structured exercise protocol targeting strength (2 days/week) and endurance (3days/week) training
  Arms: Convetional phyusical therapy

SUMMARY:
As functional electrical stimulations has evident role in improving motor control in tenodesis function (power and precision grip) but its results are considered to be short term so addition of task oriented approach i.e. motor priming exercises could enhance the treatment effects . Priming is a mechanism that could easily be a part of a restorative occupational therapy approach, is a therapeutic method with the intent to improve function by targeting underlying neural mechanisms (neuroplasticity and motor control). This will yield the long term effects of priming augmented functional electrical stimulations to enhance the tenodesis function of patients with spinal cord injury. Their combination may produce improvement in hand functions dexterity in spinal cord injury patients.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is damage to the spinal cord that causes temporary or permanent changes in or loss of muscle function, sensation, or autonomic function in the parts of the body served by the spinal cord, below the level of the injury. People with Spinal cord injury (C6-7 tetraplegia) are often lacking grip strength, causing impairment in activities of daily living. Variety of physiotherapy approaches such as electrical stimulations and different exercise regimes has been used in rehabilitation program of spinal cord injuries. Functional electrical impulses apply to nerves and muscles to restore muscle function in people with spinal cord injury. Second, priming of the motor cortex with motor priming exercises is associated with neuroplastic changes and improved motor performance.

This will be a randomized control trail and the study aims to determine which group will show better results of functional electrical stimulations with or without motor priming exercise on tenodesis grip in sub acute spinal cord injury patients. Evidences support that, in more than 40 years of functional electrical stimulation research, principles for safe stimulation of neuromuscular tissue have been established; it has been developed for restoring function in the upper extremity, lower extremity, bladder and bowel, and respiratory system. Paralyzed or paretic muscles can be made to contract by applying

electrical currents to the intact peripheral motor nerves innervating them. When electrically elicited muscle contractions are coordinated in a manner that provides function, the technique is termed functional electrical stimulation (FES)

Another approach is Motor priming, which is receiving considerable attention as a way of augmenting the effects of rehabilitation-related training in neurologic clinical populations. Much of the early work related to motor priming to improve hand function in persons with tetraplegia) Priming is a non-conscious process associated with learning where exposure to a stimulus alters the response of another stimulus. When used successfully in conjunction with a therapeutic intervention, priming results in a behavior change coinciding with changes in neural processes. Motor priming exercises demonstrate changes in cortical excitability, or facilitate cognitive processing, thus inducing neuroplastic effects such as release of neurochemicals that may enhance the effect of subsequent training. Priming that target the motor cortex is a relatively new topic of research in the fields of motor control and rehabilitation

This will be a randomized control trial and patients will be recruited through convenient sampling into three groups. Group A will be given functional electrical stimulations with motor priming exercises. Group B will be receiving functional electrical stimulations alone and group C will receive conventional exercises training. Pre and post measurements with outcome measuring tool will be taken. Tools for accessing tenodesis grip will be hand dynamometer, pinch meter, Manual Muscle Testing, graded redefined assessment of sensation , strength and pretension; GRASSP tool, Spinal Cord Independence Measure SCIM- self care sub score . The data will be analyzed using SPSS 25 software.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female with age group (15 50)
* Patient with C6-C7 neurological level of injury
* Patient with incomplete ASIA- D grading
* Clinically stable patients with normal vital signs and mental status
* Patient in acute and sub-acute stage ( usually < 18 months post injury
* Patients without active palmer and lateral grasp function (except tenodesis grasp function)
* Patients having intact wrist extensors in Grade 3 or higher manual muscle test i.e. can perform tenodesis action

Exclusion Criteria:

* Patients with Neurological level of injury C8 or above
* Patient with chronic stage > 18 months
* Patients with Spastic hands
* Patients with implants in body
* Patients with history of Epilepsy
* Patients with Cardiovascular problems

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Hand Dynamometer | 6th week
  Used to measure grip strength.The patient squeezes the dynamometer with all of their strength, typically three times with each hand. An average score is then calculated using the measurements from both hands
Pinch meter | 6th week
  A pinch meter is a medical instrument that is used to test digital strength in the form of three different types of pinches. It primarily serves as a diagnostic and assessment tool.The therapist takes the average of 3 trials for each type of pinch, alternating from one hand to the other. Positioning during the test should be shoulder adducted, elbow at 90 degrees and forearm in neutral
The American Spinal Injury Association Impairment Scale | 6th week
  The American Spinal Injury Association Impairment Scale is a standardized neurological examination used by the rehabilitation team to assess the sensory and motor levels which were affected by the spinal cord injury
Graded redefined assessment for sensation, strength and prehension tool | 6th week
  The GRASSP is a clinical impairment measure used for the upper limb after tetraplegia. The measure includes three domains (sensation, strength , prehension) which are important in describing hand function(

SECONDARY OUTCOMES:
Spinal Cord Independence Measure | 6th weeks
  The SCIM has been developed to address three specific areas of function in
  patients with spinal cord injury (SCI). It looks at self-care (feeding, grooming, bathing, and dressing), respiration and sphincter management, and a patient's mobility abilities i.e. bed mobility and transfers and indoors/outdoors

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Lahore general Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2016 Traumatic Brain Injury and Spinal Cord Injury Collaborators. Global, regional, and national burden of traumatic brain injury and spinal cord injury, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 Jan;18(1):56-87. doi: 10.1016/S1474-4422(18)30415-0. Epub 2018 Nov 26. PMID 30497965
- [Background] Jung HY, Lee J, Shin HI. The natural course of passive tenodesis grip in individuals with spinal cord injury with preserved wrist extension power but paralyzed fingers and thumbs. Spinal Cord. 2018 Sep;56(9):900-906. doi: 10.1038/s41393-018-0137-4. Epub 2018 May 22. PMID 29789707
- [Background] Peckham PH, Knutson JS. Functional electrical stimulation for neuromuscular applications. Annu Rev Biomed Eng. 2005;7:327-60. doi: 10.1146/annurev.bioeng.6.040803.140103. PMID 16004574
- [Background] Stoykov ME, Corcos DM, Madhavan S. Movement-Based Priming: Clinical Applications and Neural Mechanisms. J Mot Behav. 2017 Jan-Feb;49(1):88-97. doi: 10.1080/00222895.2016.1250716. Epub 2017 Mar 1. PMID 28277966
- [Background] Vafadar AK, Cote JN, Archambault PS. Effectiveness of functional electrical stimulation in improving clinical outcomes in the upper arm following stroke: a systematic review and meta-analysis. Biomed Res Int. 2015;2015:729768. doi: 10.1155/2015/729768. Epub 2015 Jan 22. PMID 25685805
- [Background] Sivaramakrishnan A, Madhavan S. Combining transcranial direct current stimulation with aerobic exercise to optimize cortical priming in stroke. Appl Physiol Nutr Metab. 2021 May;46(5):426-435. doi: 10.1139/apnm-2020-0677. Epub 2020 Oct 23. PMID 33095999
- [Background] Gomes-Osman J, Tibbett JA, Poe BP, Field-Fote EC. Priming for Improved Hand Strength in Persons with Chronic Tetraplegia: A Comparison of Priming-Augmented Functional Task Practice, Priming Alone, and Conventional Exercise Training. Front Neurol. 2017 Jan 17;7:242. doi: 10.3389/fneur.2016.00242. eCollection 2016. PMID 28144229
- [Background] Burns AS, Marino RJ, Kalsi-Ryan S, Middleton JW, Tetreault LA, Dettori JR, Mihalovich KE, Fehlings MG. Type and Timing of Rehabilitation Following Acute and Subacute Spinal Cord Injury: A Systematic Review. Global Spine J. 2017 Sep;7(3 Suppl):175S-194S. doi: 10.1177/2192568217703084. Epub 2017 Sep 5. PMID 29164023
- [Background] Mangold S, Keller T, Curt A, Dietz V. Transcutaneous functional electrical stimulation for grasping in subjects with cervical spinal cord injury. Spinal Cord. 2005 Jan;43(1):1-13. doi: 10.1038/sj.sc.3101644. PMID 15289804
- [Background] El Masry WS, Tsubo M, Katoh S, El Miligui YH, Khan A. Validation of the American Spinal Injury Association (ASIA) motor score and the National Acute Spinal Cord Injury Study (NASCIS) motor score. Spine (Phila Pa 1976). 1996 Mar 1;21(5):614-9. doi: 10.1097/00007632-199603010-00015. PMID 8852318
- [Background] Popovic MR, Thrasher TA, Adams ME, Takes V, Zivanovic V, Tonack MI. Functional electrical therapy: retraining grasping in spinal cord injury. Spinal Cord. 2006 Mar;44(3):143-51. doi: 10.1038/sj.sc.3101822. PMID 16130018